CLINICAL TRIAL: NCT04257344
Title: Association Between Postoperative Glucose Profile, Sleep and Heart Rate Variability and Postoperative Complications in Patients Undergoing Acute, Abdominal Surgery. A Prospective, Explorative Cohort Study
Brief Title: Use of Wearables for Early Detection of Complications After Major Acute Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-071-2019
Record Dates: First submitted 2019-12-11; First posted 2020-02-06 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Surgery--Complications; Abdomen Disease
Keywords: Wearables; Emergency surgery; Abdominal surgery; Patient reported outcome measures; Recovery; Continues Glucose Monitoring; Heart Rate Variation; Actigraphy; Sleep; Quality of Recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to investigate whether glucose profile, sleep disturbances and heart rate variability measured with wearable devices is associated with postoperative recovery and complications within 30 days after major emergency abdominal surgery.

The study is designed as an explorative, prospective cohort study. 40 patients undergoing major emergency abdominal surgery at Zealand's University Hospital Køge are included in the study, and inclusion occurs within 24 hours of end of surgery. Patients will be followed for 30 days, and three scheduled study visits are planned during follow up at postoperative day 10, 20 and 30.

Glucose is measured continuously with a wearable subcutaneous sensor (Dexcom G6). Glucose readings are validated in the perioperative setting using blood glucose measurements obtained with standard finger-pricks 3-5 times a day during hospitalization.

Actigraphy is used for assessing sleep- and activity patterns for the full study period.

Heart rate variation is measured with a compact Holter monitor. Furthermore, the study assesses patient-reported quality of recovery, glucose metabolism, nutritional status and mobility. Various data on demographics, peri- and postoperative data will be extracted from the electronic patient chart.

DETAILED DESCRIPTION:
Purpose:

The purpose of the study is to investigate the glucose-profile, HRV and sleep disturbances for 30 days after major emergency abdominal surgery using continues measurements with wearable devices. Secondly, the study investigates the association between glucose profile, HRV, sleep-disturbances, patient reported recovery and postoperative complications.

Design and study population:

The study is designed as a prospective, explorative cohort study applying repeated measures. Patients undergoing major emergency abdominal surgery at Zealand's University Hospital Køge are included. Included patients receive a standardized treatment regimen (Optimizing Major EmerGency Abdominal surgery, OMEGA), which has been established in the surgical department in order to reduce unnecessary waiting time and optimize and standardize treatment before, during and after major emergency abdominal surgery. The treatment regimen includes pre-operative antibiotics, I.V. fluid, pain and nausea treatment, nasogastric tube and prioritized, fast access to CT-scans and final surgical treatment.

Sample Size:

To the extent of our knowledge, no prior studies have simultaneously investigated sleep disturbances, heart rate variability and glucose profile using continues measurements with wearables before and up to 30 days after major emergency abdominal surgery. A traditional power calculation would be based on arbitrary data and is therefore omitted. Hence, the present study is designed as an exploratory study with no primary endpoint and functions as a pilot study prior to future larger, focused cohort studies. It is estimated, that inclusion of 40 patients in the present study is feasible and provides sufficient statistical power to show significant changes and association between glucose profile, HRV, sleep patterns and patient reported outcome measures.

Course of the study and assessment tools:

Eligible patients will be contacted by study investigators within 12-24 hours after surgery when the patient has been re-transferred to the surgical ward. Included patients will be followed for 30 days, and three scheduled study visits are planned during follow up at postoperative day 10, 20 and 30.

Glucose is measured continuously from the interstitial fluid of the subcutaneous tissue with a wearable subcutaneous sensor (Dexcom G6). Continues Glucose measurement (CGM) is normally used by diabetic patients in an outpatient setting. Therefore, the CGM readings are validated in the perioperative setting using capillary blood glucose measurements obtained with standard finger-pricks 3-5 times a day during hospitalization. The CGM-monitor is mounted on the patient from inclusion until 30 days after surgery. Metrics of within-day glycemic variability include the standard deviation (SD), the 'mean amplitude of glucose excursions' (MAGE) and the 'derived coefficient of variation' (%CV). Stable glucose levels are defined as a %CV <36% according to the international consensus on use of continues glucose monitoring. Metrics of between-day glucose variability include 'Mean of daily differences' (MODD), which is the absolute difference between two glucose values measured at the same time with a 24 h interval. Furthermore, the daily 'mean glucose level' and 'time in ranges' (TIRs) will be reported.

Actigraphy is used for measuring sleep- and activity patterns for the full study period. The device consists of three linear accelerometer with an integrated minicomputer that allows the direct measure of accelerations in all directions. In this study we will use the 'Zero-crossing method', where every acceleration (>0,1g) during each epoch length are measured. The epoch length in this study is predefined to 60 seconds. Metrics of sleep disturbances include 'Time in Bed' (TIB), 'Total Sleep Time' (TST), ' Sleep Efficiency' (SE), 'Wake Time' (WT) and 'Wake after Sleep Onset' (WASO), Sleep Latency (SL) and number of awakenings longer than five minutes" (NOA).

A battery powered, rechargeable heart rate monitor (C3 Holter monitor, Cortrium, Denmark) will be used for monitoring HRV. The device is a triangular monitor (7x7x7cm) and consist of three integrated electrodes allowing for measuring long term ECG. Data is stored on internal memory on the device and can be transferred to appropriate desktop software (Kubios Premium). Heart rate will be monitored from inclusion until 7 days after discharge or until postoperative day 14, whatever comes first. Time-domain analysis of HRV will be applied as recommended in the guidelines from the European Society of Cardiology and The North American Society of Pacing and Electrophysiology.

The widely used questionnaire quality of recovery-15 (QoR/15) quantifies patient reported quality of recovery with 15 Danish translated and validated questions. The questionnaire is completed in 2-3 minutes and results in a score up to 150 points with a high score indicating high self-reported postoperative recovery. The participants fills out QoR-15 every day during hospitalization and once at each scheduled study visit.

Estimation of pancreatic beta-cell functions and peripheral insulin resistance will be assessed with paired C-peptide and plasma glucose samples obtained at inclusion, discharge and 30-day follow up. In addition, changes in p-carbamide, hemoglobin, hemoglobin A1C, C-reactive protein and white blood cell count are measured during the study period.

A designated dietician assesses the patient's daily nutritional energy intake during hospitalization. In addition, the patient's nutritional consumption after discharge is estimated with the "24 hour recall method" at each follow up visit and the questionnaire "Food Frequency questionnaire" (FFQ), at 30 day follow up. In the FFQ-questionnaire, the patient reports the frequency of the consumption of 104 different common food and drink products during the last 30 days.

To assess changes in the patient's mobility the "Timed Up-and-go"-test will be used. Furthermore, 7 basic abilities during hospitalization (e.g. showering or dressing) are assessed on a scale from 0-2 with the questionnaire "Mobility during Hospitalization". After discharge, the questionnaire "Activity of Daily Living (ADL)" is used for assessing whether the patient is able to perform everyday activities (e.g. cooking, grossery shopping) on a 1-5 scale. In addition, handgrip strength, weight and bio impendence is measured at inclusion, at discharge and at each follow up visit.

Data on demographics, peri- and postoperative data will be extracted from the electronic patient chart. Postoperative complications will be classified according to the Clavien-Dindo classification.

To investigate the subjective experience of being discharged with three wearable monitors, a designated anthropologist conducts a semi-structured interview in a subgroup of 6-8 patients.

Statistics:

For baseline characteristics, descriptive statistics will be applied including reports of mean, standard deviation (SD), median and interquartile range (IQR) when appropriate. For comparison, chi^2 test and t-test will be applied. When data is not normally distributed, log-transformation will be used when possible. Further statistical methods include correlation analysis and logistic regression modelling with adjustment of relevant confounders. A two-tailed p-value of 0.05 is considered statistically significant. Designated statistical software will be used (e.g. R version 3.6.1, https://www.r-project.org/). A trained statistician will be consulted when analyzing data.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major emergency abdominal surgery including laparotomy or laporoscopy. Indications include ileus, perforated hollow organ, intraabdominal bleeding, ischemia, wound dehiscence.

Exclusion Criteria:

* Laparoscopic surgeries for diseases related to appendix, gall bladder or bile ducts are excluded, unless the procedure is converted to open surgery perioperative.
* not understanding or speeking danish
* cognitive dysfunction
* chronic immobilization
* pregnancy
* diabetes (type I and II)
* Permanent atrial fibrillation or pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population consists of all patients admitted at Zealands University Hospital Køge, who undergo major emergency abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-15 score | 30 days
  The score is based on 15 questions with a maximum total score of 150 indicating excellent patient-reported recovery
Heart rate variation | 7 days post discharge or maximum 14 days after surgery
  Heart rate variation measured with wearable devices. Time domain measures are used.
Total Sleep Time | 30 days
  Total time of sleep during 24 hours, assessed with actigraphy
Sleep Efficiency | 30 days
  The ratio of the total sleep time compared to the total time spent in bed during 24 hours
Mean amplitude of glucose excursions (MAGE) | 30 days
  Measure of within-day glycemic variability assessed with continues glucose monitoring

SECONDARY OUTCOMES:
Time in bed | 30 days
  total time in bed during 24 hours, assessed with actigraphy
Wake Time | 30 days
  Time awake during 24 hours assessed with acitgraphy
Wake after Sleep Onset (WASO) | 30 days
  Total time awake after sleep onset assessed with actigraphy
Number of awakenings | 30 days
  Number of awakenings longer than five minutes assessed with actigraphy
Time in range | 30 days
  The total time during 24 hours where the patient is normoglycemic, assessed with continues glucose monitoring
Mean glucose level | 30 days
  The mean glucose level during 24 hours assessed with continues glucose monitoring
Derived coefficient of glucose variation (%CV) | 30 days
  Measure of within-day glycemic variability

CONTACTS AND LOCATIONS:
Overall Officials: Johan Johan, MD, Principal Investigator — Surgical department, Zealands University Hospital
Locations (1):
- Surgical department, Zealand University Hospital, Køge, Denmark

REFERENCES:
- [Background] Monnier L, Colette C, Owens DR. The application of simple metrics in the assessment of glycaemic variability. Diabetes Metab. 2018 Sep;44(4):313-319. doi: 10.1016/j.diabet.2018.02.008. Epub 2018 Mar 6. PMID 29602622
- [Background] Danne T, Nimri R, Battelino T, Bergenstal RM, Close KL, DeVries JH, Garg S, Heinemann L, Hirsch I, Amiel SA, Beck R, Bosi E, Buckingham B, Cobelli C, Dassau E, Doyle FJ 3rd, Heller S, Hovorka R, Jia W, Jones T, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Maahs D, Murphy HR, Norgaard K, Parkin CG, Renard E, Saboo B, Scharf M, Tamborlane WV, Weinzimer SA, Phillip M. International Consensus on Use of Continuous Glucose Monitoring. Diabetes Care. 2017 Dec;40(12):1631-1640. doi: 10.2337/dc17-1600. PMID 29162583
- [Background] Berger AM, Wielgus KK, Young-McCaughan S, Fischer P, Farr L, Lee KA. Methodological challenges when using actigraphy in research. J Pain Symptom Manage. 2008 Aug;36(2):191-9. doi: 10.1016/j.jpainsymman.2007.10.008. Epub 2008 Apr 8. PMID 18400460
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Wallace TM, Levy JC, Matthews DR. Use and abuse of HOMA modeling. Diabetes Care. 2004 Jun;27(6):1487-95. doi: 10.2337/diacare.27.6.1487. PMID 15161807
- [Background] Beer-Borst S, Amado R. Validation of a self-administered 24-hour recall questionnaire used in a large-scale dietary survey. Z Ernahrungswiss. 1995 Sep;34(3):183-9. doi: 10.1007/BF01623156. PMID 7502539
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946